CLINICAL TRIAL: NCT04496011
Title: Effect of the Use of a Cycloergometer on the Physical Performance of Patients Undergoing Hematopoietic Stem Cell Transplantation: A Randomized and Controlled Clinical Trial
Brief Title: Effect of the Cycloergometer in Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, Sponsor-Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TMO 2020
Record Dates: First submitted 2020-06-07; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Fatigue; Leukemia; Lymphoma; Multiple Myeloma; Hematopoietic Stem Cell Transplantation
Keywords: Autologous transplant; Allogeneic transplant; Physiotherapy; Exercise; Fatigue
MeSH Terms: conditions — Fatigue; Leukemia; Lymphoma; Multiple Myeloma; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will be included by convenience (according to the inclusion and exclusion criteria) in non-probabilistic form. The included individuals will be randomized by (nome do Sofwate) in two lists: one for the control group and other for the experimental group. Once defined that the patient will be part of the experimental group, a bicycle ergometer will be kept in the patient's accommodation during the period of hospitalization due to restrictions imposed by the Infection Control Department. Thus, the equipment will remain in the patient´s room during the hospitalization, while the other patients will be allocated to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In this group the exercise program will be based on the protocol of Control Group, without the exception of walking training, adding aerobic capacity training using the bicycle ergometer, model CBL11 Classic® from ACT®.
  Interventions: Other: Aerobic training with cycle ergometer
- Group Control (No Intervention): In this group the exercise program is based on the standard physiotherapy protocol that is part of the care routines performed at the bone marrow transplant service.
  It includes essential components of a rehabilitation program: range of motion, balance training, gait and strength of the upper and lower limbs

INTERVENTIONS:
Other: Aerobic training with cycle ergometer — Patients start with an initial warm-up of 2 minutes, with rotations per minute free, without load. Progressively, the load of the exercise cycle increases every minute up to the supported limit or up to 60% - 70% of maximum heart rate (HRmax). The training will be carried out for 20 continuous minutes, being interrupted whenever the heart rate (HR) reaches 90% of the maximum expected for the age and / or the loss of effort perceived in the BORG scale, above 8 on a scale of 0 to 10.
  Arms: Experimental Group

SUMMARY:
Physiological changes caused by hematological diseases associated with high dose chemotherapy have a negative impact on patient's functionality, making them more fragile and vulnerable after hematopoietic cell transplantation. Currently, randomized studies have shown that physical exercise can contribute to improve Quality of Life of these patients. In this randomized controlled trial, we will study the effect of using the bicycle ergometer on the physical performance of patients undergoing transplantation of hematopoietic stem cells (HSCT).

DETAILED DESCRIPTION:
The sample consists of 30 patients diagnosed with leukemia, lymphoma and multiple myeloma, undergoing high-dose chemotherapy and hematopoietic stem cells transplantation, who will be randomized into two groups. The results of muscle strength in the lower limbs, general mobility, fatigue and clinical symptoms will be compared between the control group and the experimental group.

The control group will perform an exercise program based on the standard protocol of the physiotherapy service, where exercises are performed to gain strength in muscle groups of the upper and lower limbs, range of motion, balance and functional movements. The experimental group will perform the same exercises as the control group, added to a training program using a bicycle ergometer, with an incremental load (from 60% to 70% of the maximum heart rate) for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-70 years) scheduled to perform the first HSCT;
* Be with a preserved neurological function and full cognition;
* Have clinical conditions that allow participation in the motor physiotherapy program;
* Be agreed with a study proposal and sign the free and informed consent form (ICF).

Exclusion Criteria:

* Develop clinical complications that contraindicate the performance of motor physiotherapy including the practice of the cycle ergometer;
* Present a previous musculoskeletal alteration that interferes with the performance of physical performance assessment tests;
* Recent cardiovascular or pulmonary disease;
* Psychiatric or neurological disorder;
* Need for gait assistance or presence of bone metastasis
* Adherence below 50% of the total motor physiotherapy protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Lower Limb Physical Functioning and Strength | Trough study completion, an average of 2 months
  The 30-Second Chair Stand evaluates lower limb strength and, indirectly, the risk of falls, especially in the elderly population (JONES, J., RIKLI, 2002). This way, it will compose the set of tests used to determine the physical performance by measuring the number of stands from an armless chair of standard height (45 cm) performed in 30 seconds. The test will be begin when the participant, seating on a neutral spine position and feet flat on the floor, will be instructed to rise to a full stand and return to the original seated position, as quickly as possible. The participant will be instructed to move at maximal speed until they either feel the need to stop or the 30-second time limit is reached. More than 8 unassisted stands for men and women are considered above average for their age, and those below the range as below average

SECONDARY OUTCOMES:
Fatigue | Trough study completion, an average of 2 months
  Piper Fatigue Scale, developed by Piper et al. (1998), is a multidimensional measure of fatigue in the field of cancer research and includes subdomains of the behavioral, affective, sensorial and cognitive attributes / fatigue mood, composed of 22 items. The scores for each item range from 0 to 10 and can total 220 points. Higher values characterize a greater perception of fatigue. It will be applied on patient's evaluation day and on hospital discharge day.
Symptoms Assessment | Trough study completion, an average of 2 months
  The Edmonton Symptom Assessment Scalemorning will be applied to eavaluate symptoms of pain, tiredness, drowsiness, appetite, nausea, shortness of breath, depression, anxiety and well-being. It is a scale where the patient provides an auto-report on a score that can vary from 0 to 10, being score 0 absence of symptoms and 10 represents the most intense sensation experienced by the patient.
Timed up and Go (TUG) | Trough study completion, an average of 2 months
  TUG is used in clinical practice to assess mobility, the risk of falls and also to assist in the diagnosis of sarcopenia. For this reason, that test will be compiled or set of tests that will be used to determine physical performance.

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio Edler Macagnan, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre - UFCSPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No